CLINICAL TRIAL: NCT02775149
Title: Dental Erosion in Patients With Gastro-oesophageal Reflux
Status: Suspended | Type: Observational
Why Stopped: No participants
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Philipp Kanzow, Dr. med. dent., Dr. rer. medic., Dr. med. dent., University Medical Center Goettingen
Other Study IDs: Erosion-Reflux; 2/11/15 (Other: Ethics Committee of the University Medical Center Göttingen)
Record Dates: First submitted 2016-05-09; First posted 2016-05-17 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Dental Erosion
MeSH Terms: conditions — Tooth Erosion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples are obtained and retained for 10 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Reflux patients: Patients who are treated at the Clinic for Gastroenterology and Gastrointestinal Oncology and have a 24-hours pH monitoring or impedance measurement performed for medical reasons
  Interventions: Other: Collection of saliva samples; Other: Visual detection of BEWE-index

INTERVENTIONS:
Other: Collection of saliva samples — Collection of saliva samples
Other: Visual detection of BEWE-index — Visual detection of BEWE-index

SUMMARY:
Not only caries but also exposure to acids can lead to loss of tooth structure. This acid-related tooth structure loss is defined as dental erosion.

A relationship between dental erosion and occurence of reflux disease was shown in numerous studies. On the one hand, patients with dental erosions frequently show reflux disease. On the other hand, many - but not all - reflux patients show dental erosions. It is believed that certain salivary parameters might explain, why not all reflux patients alike are affected of dental erosions.

The aim of this study is to analyze the relationship and the extent of occurrence of dental erosions and reflux symptoms, including investigation of certain salivary parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are treated at the Clinic for Gastroenterology and Gastrointestinal Oncology and have a 24-hours pH monitoring or impedance measurement performed for medical reasons

Exclusion Criteria:

* Inability to give written consent
* Age <18 years
* Intake of proton pump inhibitors (PPIs) if they are not discontinued at least one week before study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Exploratory study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Visual assessment of the BEWE-(basic erosive wear examination)-index | After removal of the probe (on second day)

SECONDARY OUTCOMES:
Determination of unstimulated and stimulated saliva flow rate (ml/min). | While wearing the probe at three time points over 24h: morning, noon, evening
Determination of saliva pH and buffer capacity (mol/L). | While wearing the probe at three time points over 24h: morning, noon, evening
Determination of total protein content in saliva (g/L). | While wearing the probe at three time points over 24h: morning, noon, evening
Determination inorganic calcium and phosphate in saliva (mmol/L). | While wearing the probe at three time points over 24h: morning, noon, evening
Measurement of salivary enzyme activity: Protease, Kollagenase/Gelatinase, Pepsin, Trypsin, and Amylase (U/mL). | While wearing the probe at three time points over 24h: morning, noon, evening

CONTACTS AND LOCATIONS:
Overall Officials: Annette Wiegand, Prof. Dr. med. dent., Principal Investigator — Dept. of Prev. Dentistry, Periodontology and Cariology, University Medical Center Göttingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartlett D, Ganss C, Lussi A. Basic Erosive Wear Examination (BEWE): a new scoring system for scientific and clinical needs. Clin Oral Investig. 2008 Mar;12 Suppl 1(Suppl 1):S65-8. doi: 10.1007/s00784-007-0181-5. Epub 2008 Jan 29. PMID 18228057
- [Background] Hara AT, Zero DT. The potential of saliva in protecting against dental erosion. Monogr Oral Sci. 2014;25:197-205. doi: 10.1159/000360372. Epub 2014 Jun 26. PMID 24993267
- [Background] Moazzez R, Bartlett D, Anggiansah A. Dental erosion, gastro-oesophageal reflux disease and saliva: how are they related? J Dent. 2004 Aug;32(6):489-94. doi: 10.1016/j.jdent.2004.03.004. PMID 15240067
- [Background] Ranjitkar S, Smales RJ, Kaidonis JA. Oral manifestations of gastroesophageal reflux disease. J Gastroenterol Hepatol. 2012 Jan;27(1):21-7. doi: 10.1111/j.1440-1746.2011.06945.x. PMID 22004279
- [Background] Schlueter N, Ganss C, Potschke S, Klimek J, Hannig C. Enzyme activities in the oral fluids of patients suffering from bulimia: a controlled clinical trial. Caries Res. 2012;46(2):130-9. doi: 10.1159/000337105. Epub 2012 Apr 3. PMID 22472533
- [Background] Wang GR, Zhang H, Wang ZG, Jiang GS, Guo CH. Relationship between dental erosion and respiratory symptoms in patients with gastro-oesophageal reflux disease. J Dent. 2010 Nov;38(11):892-8. doi: 10.1016/j.jdent.2010.08.001. Epub 2010 Aug 7. PMID 20696201
- [Background] Wilder-Smith CH, Materna A, Martig L, Lussi A. Gastro-oesophageal reflux is common in oligosymptomatic patients with dental erosion: A pH-impedance and endoscopic study. United European Gastroenterol J. 2015 Apr;3(2):174-81. doi: 10.1177/2050640614550852. PMID 25922678
- [Background] Kanzow P, Wegehaupt FJ, Attin T, Wiegand A. Etiology and pathogenesis of dental erosion. Quintessence Int. 2016 Apr;47(4):275-8. doi: 10.3290/j.qi.a35625. PMID 27022647